CLINICAL TRIAL: NCT07095907
Title: Post-surgical Functional Results in Patients With Epiretinal Membrane Undergoing Controlled Macular Detachment: Pilot Study.
Brief Title: Post-surgical Functional Results in Patients With Epiretinal Membrane Undergoing Controlled Macular Detachment
Acronym: DMER25
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RE-25-09
Record Dates: First submitted 2025-07-09; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Epiretinal Membrane Surgery
Keywords: Epiretinal membrane; Epiretinal membrane surgery; Macular detachment
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Intervention Model Description: Prospective, Longitudinal, Experimental, Descriptive Cohort Study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient protocol (Experimental): Patients over 18 years of age, with a clinical diagnosis of Epiretinal Membrane grade 3 and 4 according to Optical Coherence Tomography, who attend the Retina service.
  Interventions: Procedure: Pars plana vitrectomy with epiretinal membrane peeling and controlled macular detachment

INTERVENTIONS:
Procedure: Pars plana vitrectomy with epiretinal membrane peeling and controlled macular detachment — Currently, vitrectomy with epiretinal membrane peeling is the standard procedure; however, its ability to improve visual acuity in these patients remains limited. In this context, controlled macular detachment is emerging as a surgical alternative that could optimize the anatomical and functional restoration of the retina.

SUMMARY:
This study aims to evaluate postsurgical functional changes in patients with advanced epiretinal membrane (ERM) (stages 3 and 4) by integrating a controlled macular detachment with a balanced salt solution to the conventional ERM peeling technique.

DETAILED DESCRIPTION:
The evolution of visual acuity will be analyzed using the ETDRS letter scale. At the same time, anatomical and microvascular changes will be evaluated using optical coherence tomography (OCT) and optical coherence tomography angiography (OCT-A) to evaluate their impact on visual recovery. This technique is expected to minimize persistent distortion, promote restoration of retinal perfusion, mitigate postoperative ischemia, and improve macular structural stability, potentially leading to more significant functional recovery. It is designed as a prospective longitudinal pilot study; The research will be carried out in the Retina Department of the Association to Prevent Blindness in Mexico (APEC), focusing on patients over 18 years of age with a diagnosis of advanced MRD and eligible for vitreoretinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with a confirmed diagnosis of ERM grade III or IV by Optical Coherence Tomography who present visual disturbances such as metamorphopsia or visual impairment (measured in letters on the ETDRS scale) but who do not reflect end-stage visual impairment.
* Patients suitable for vitreoretinal surgical procedures, with no uncontrolled medical comorbidities that contraindicate surgery.
* Patients who understand the objectives and risks of the study and sign an informed consent form.

Exclusion Criteria:

* Patients with a confirmed diagnosis of grade III or IV ERM by Optical Coherence Tomography who do not have the ability to improve their visual acuity.
* Patients diagnosed with ocular pathologies that significantly affect their visual acuity, such as moderate or advanced glaucoma, non-glaucomatous optic neuropathies, or optic media opacities such as leukomas, significant corneal edema, or other maculopathies such as macular atrophy or macular ischemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-12-17 (Estimated); Study Completion 2026-01-26 (Estimated)

PRIMARY OUTCOMES:
BCVA (Best corrected visual acuity) | From the first recruitment evaluation to the last one at 3 months post-surgery
  Ability to discriminate fine details at a standard distance, assessed by reading letters on an ETDRS chart.

SECONDARY OUTCOMES:
Postoperative anatomical changes of the macula using optical coherence tomography: Central macular thickness (µm) | From enrollment to the end of follow-up at the third month.
  Central macular thickness measured in microns (µm)
Postoperative anatomical changes of the macula using optical coherence tomography: Inner nuclear layer thickness (µm) | From enrollment to the end of follow-up at the third month.
  Inner nuclear layer thickness measured in microns (µm)
Postoperative anatomical changes of the macula using optical coherence tomography: Ellipsoid zone disruption | From enrollment to the end of follow-up at the third month.
  Presence or absence of disruption of the Ellipsoid layer

CONTACTS AND LOCATIONS:
Overall Officials: Raul Velez, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Hospital Asociación Para Evitar la Ceguera en México I.A.P., Mexico City, Mexico

REFERENCES:
- [Background] Abu-Ain M, Shatnawi R, Shehadeh I, Khan MI. Long-Term Visual Acuity and Optical Coherence Tomography Changes After Vitrectomy for Idiopathic Epiretinal Membranes. Clin Ophthalmol. 2023 Feb 28;17:693-700. doi: 10.2147/OPTH.S401017. eCollection 2023. PMID 36880022
- [Background] Chang WC, Lin C, Lee CH, Sung TL, Tung TH, Liu JH. Vitrectomy with or without internal limiting membrane peeling for idiopathic epiretinal membrane: A meta-analysis. PLoS One. 2017 Jun 16;12(6):e0179105. doi: 10.1371/journal.pone.0179105. eCollection 2017. PMID 28622372
- [Background] Khanna RK, Dorvault M, Pasco J, Cook AR, Pichard T, Marotte MT, Pisella PJ, Arsene S. Long-term functional outcomes and vision-related quality of life after vitrectomy for epiretinal membrane: a prospective cohort study. Sci Rep. 2022 Feb 15;12(1):2470. doi: 10.1038/s41598-022-06482-3. PMID 35169203
- [Background] Flaxel CJ, Adelman RA, Bailey ST, Fawzi A, Lim JI, Vemulakonda GA, Ying GS. Idiopathic Epiretinal Membrane and Vitreomacular Traction Preferred Practice Pattern(R). Ophthalmology. 2020 Feb;127(2):P145-P183. doi: 10.1016/j.ophtha.2019.09.022. Epub 2019 Sep 25. No abstract available. PMID 31757497
- [Background] Morizane Y, Kimura S, Hosokawa M, Shiode Y, Hirano M, Doi S, Hosogi M, Fujiwara A, Inoue Y, Shiraga F. Planned foveal detachment technique for the resolution of diffuse diabetic macular edema. Jpn J Ophthalmol. 2015 Sep;59(5):279-87. doi: 10.1007/s10384-015-0390-4. Epub 2015 Jul 30. PMID 26220819
- [Background] Szurman P, Roters S, Grisanti S, Aisenbrey S, Schraermeyer U, Luke M, Bartz-Schmidt KU, Thumann G. Ultrastructural changes after artificial retinal detachment with modified retinal adhesion. Invest Ophthalmol Vis Sci. 2006 Nov;47(11):4983-9. doi: 10.1167/iovs.06-0491. PMID 17065517
- [Background] Momota A, Iwase T, Akahori T, Goto K, Yamamoto K, Ra E, Terasaki H. Association between displacement and thickness of macula after vitrectomy in eyes with epiretinal membrane. Sci Rep. 2020 Aug 6;10(1):13227. doi: 10.1038/s41598-020-70197-6. PMID 32764657
- [Background] Choi KE, Kim S, Kim SW. Anatomical changes in idiopathic epiretinal membrane at 2-year follow-up assessed using spectral domain optical coherence tomography and optical coherence tomographic angiography. Graefes Arch Clin Exp Ophthalmol. 2024 May;262(5):1465-1474. doi: 10.1007/s00417-023-06332-6. Epub 2023 Dec 20. PMID 38117309
- [Background] Bacherini D, Dragotto F, Caporossi T, Lenzetti C, Finocchio L, Savastano A, Savastano MC, Barca F, Dragotto M, Vannozzi L, Nasini F, Faraldi F, Rizzo S, Virgili G, Giansanti F. The Role of OCT Angiography in the Assessment of Epiretinal Macular Membrane. J Ophthalmol. 2021 Mar 24;2021:8866407. doi: 10.1155/2021/8866407. eCollection 2021. PMID 33815835
- [Background] Baldascino A, Carla MM, Vielmo L, Gambini G, Marzano FC, Margollicci F, D'Onofrio NC, Rizzo S. Microvascular Changes after Epiretinal Membrane Vitrectomy with Intraoperative Intravitreal Dexamethasone Implant: An OCT Angiography Analysis. Diagnostics (Basel). 2024 Feb 13;14(4):411. doi: 10.3390/diagnostics14040411. PMID 38396450
- [Background] Wong R, Howard C, Orobona GD. RETINA EXPANSION TECHNIQUE FOR MACULAR HOLE APPOSITION REPORT 2: Efficacy, Closure Rate, and Risks of a Macular Detachment Technique to Close Large Full-Thickness Macular Holes. Retina. 2018 Apr;38(4):660-663. doi: 10.1097/IAE.0000000000001705. PMID 28816729
- [Background] Yang HS, Choi S, Kim S, Min CH, Kim D, Lee Y, Kim M, Koo D, Ryu J, Kim J. Epiretinal Membrane: Correlations Among Clinical, Immunohistochemical, and Biochemical Features and Their Prognostic Implications. Invest Ophthalmol Vis Sci. 2024 Dec 2;65(14):25. doi: 10.1167/iovs.65.14.25. PMID 39661356
- [Background] Miyazato M, Iwashita Y, Hirono K, Ching J, Nakamura K, Inoue T, Asaoka R, Yanagi Y, Maruyama-Inoue M, Kadonosono K. Predictive factors for postoperative visual function in eyes with epiretinal membrane. Sci Rep. 2023 Dec 14;13(1):22198. doi: 10.1038/s41598-023-49689-8. PMID 38097656
- [Background] Govetto A, Virgili G, Rodriguez FJ, Figueroa MS, Sarraf D, Hubschman JP. FUNCTIONAL AND ANATOMICAL SIGNIFICANCE OF THE ECTOPIC INNER FOVEAL LAYERS IN EYES WITH IDIOPATHIC EPIRETINAL MEMBRANES: Surgical Results at 12 Months. Retina. 2019 Feb;39(2):347-357. doi: 10.1097/IAE.0000000000001940. PMID 29160787
- [Background] Govetto A, Lalane RA 3rd, Sarraf D, Figueroa MS, Hubschman JP. Insights Into Epiretinal Membranes: Presence of Ectopic Inner Foveal Layers and a New Optical Coherence Tomography Staging Scheme. Am J Ophthalmol. 2017 Mar;175:99-113. doi: 10.1016/j.ajo.2016.12.006. Epub 2016 Dec 18. PMID 27993592
- [Background] Wiznia RA. Posterior vitreous detachment and idiopathic preretinal macular gliosis. Am J Ophthalmol. 1986 Aug 15;102(2):196-8. doi: 10.1016/0002-9394(86)90144-3. PMID 3740180
- [Background] Joshi M, Agrawal S, Christoforidis JB. Inflammatory mechanisms of idiopathic epiretinal membrane formation. Mediators Inflamm. 2013;2013:192582. doi: 10.1155/2013/192582. Epub 2013 Nov 11. PMID 24324293
- [Background] Hikichi T, Takahashi M, Trempe CL, Schepens CL. Relationship between premacular cortical vitreous defects and idiopathic premacular fibrosis. Retina. 1995;15(5):413-6. doi: 10.1097/00006982-199515050-00007. PMID 8594634
- [Background] Liew G, Nguyen H, Ho IV, White AJ, Burlutsky G, Gopinath B, Mitchell P. Prevalence of Vitreoretinal Interface Disorders in an Australian Population: The Blue Mountains Eye Study. Ophthalmol Sci. 2021 Apr 19;1(2):100019. doi: 10.1016/j.xops.2021.100019. eCollection 2021 Jun. PMID 36249297
- [Background] Karasavvidou EM, Panos GD, Koronis S, Kozobolis VP, Tranos PG. Optical coherence tomography biomarkers for visual acuity in patients with idiopathic epiretinal membrane. Eur J Ophthalmol. 2021 Nov;31(6):3203-3213. doi: 10.1177/1120672120980951. Epub 2020 Dec 14. PMID 33307784
- [Background] Aung KZ, Makeyeva G, Adams MK, Chong EW, Busija L, Giles GG, English DR, Hopper J, Baird PN, Guymer RH, Robman LD. The prevalence and risk factors of epiretinal membranes: the Melbourne Collaborative Cohort Study. Retina. 2013 May;33(5):1026-34. doi: 10.1097/IAE.0b013e3182733f25. PMID 23400080
- [Background] Fung AT, Galvin J, Tran T. Epiretinal membrane: A review. Clin Exp Ophthalmol. 2021 Apr;49(3):289-308. doi: 10.1111/ceo.13914. Epub 2021 Mar 24. PMID 33656784

DOCUMENTS (1):
  • Study Protocol (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07095907/Prot_000.pdf